CLINICAL TRIAL: NCT00718484
Title: A Phase II Multicenter, Parallel Group, Randomized Study of Palifosfamide Tris Plus Doxorubicin Versus Doxorubicin in Subjects With Unresectable or Metastatic Soft-tissue Sarcoma
Brief Title: A Study of Palifosfamide Tris Plus Doxorubicin Versus Doxorubicin in Unresectable or Metastatic Soft-tissue Sarcoma
Acronym: PICASSO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IPM2002
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Soft Tissue Sarcoma
Keywords: Sarcoma; Soft Tissue Sarcoma; Doxorubicin; anthracyclin; Palifosfamide; IFOS
MeSH Terms: conditions — Sarcoma | interventions — Ifosfamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): On Day 1 of each cycle (21 days), 150 mg/m2 IV (intravenous) palifosfamide tris and 75 mg/m2 IV doxorubicin are administered on the same day. Doxorubicin administration will be initiated approximately 60 minutes after the completion of palifosfamide tris dosing. Palifosfamide tris alone is administered on Days 2 and 3, every 3 weeks (one 21-day cycle).
  Interventions: Drug: Palifosfamide Tris and Doxorubicin
- B (Active Comparator): On Day 1 of each cycle, 75 mg/m2 doxorubicin is administered IV.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Palifosfamide Tris and Doxorubicin — On Day 1 of each cycle (21 days), 150 mg/m2 IV (intravenous) palifosfamide tris and 75 mg/m2 IV doxorubicin are administered on the same day. Doxorubicin administration will be initiated approximately 60 minutes after the completion of palifosfamide tris dosing. Palifosfamide tris alone is administered on Days 2 and 3, every 3 weeks (one 21-day cycle).
  Arms: A
Drug: Doxorubicin — On Day 1 of each cycle, 75 mg/m2 doxorubicin is administered IV.
  Arms: B

SUMMARY:
This is a randomized, controlled trial to evaluate the clinical benefit of palifosfamide tris administered with doxorubicin in combination, compared with single-agent doxorubicin administered in subjects diagnosed with unresectable or metastatic soft-tissue sarcoma (STS). Subjects who meet the entry criteria will be randomized into 1 of 2 arms: either to receive palifosfamide tris plus doxorubicin or treatment with single-agent doxorubicin. Subjects will be anthracyclin naïve.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Histological or cytological documentation of sarcoma (excluding alveolar soft-part sarcoma, chondrosarcoma, dermatofibrosarcoma, Ewing sarcoma, GIST, Kaposi sarcoma, mixed mesodermal tumor, osteosarcoma, radiation induced sarcomas, and unresectable low grade liposarcoma) who have failed ≤2 prior regimens including adjuvant therapy, or ≤1 prior regimen for metastatic/unresectable disease, and for whom treatment with doxorubicin is considered medically acceptable. Prior treatment with IFOS is acceptable.
3. Have measurable disease as per RECIST criteria (Appendix 2)
4. ECOG Performance Status of 0 or 1 (Appendix 3)
5. Anthracyclin naïve
6. Life expectancy of ≥12 weeks
7. Adequate bone marrow, liver, and renal function, as assessed by the following laboratory requirements conducted within 14 days prior to dosing:

   1. Hemoglobin ≥9.0 g/dL
   2. Absolute neutrophil count (ANC) ≥1,500/mm3
   3. Platelet count 100,000/mm3
   4. Total bilirubin ≤1.5×ULN (upper limit of normal)
   5. ALT and AST ≤2.5×ULN or 5×ULN with hepatic disease
   6. Partial thromboplastin [PT]-INR/activated partial thromboplastin time [PTT] <1.5×ULN (≤2.0×ULN for subjects on anticoagulation prophylactic regimen). Subjects who are being therapeutically anticoagulated with an agent such as Coumadin (warfarin sodium) or heparin are allowed provided there is no prior evidence of underlying abnormality in coagulation parameters. If an interaction between study drug and anticoagulant is suspected, anticoagulation monitoring should be increased as appropriate.
   7. Serum creatinine ≤ULN
8. Written informed consent must be obtained from a potential subject prior to the conduct of any study-specific procedures
9. Male and female subjects must agree to use adequate birth control measures/barrier control during the course of the trial
10. Women of childbearing potential must have a urine pregnancy test performed within 14 days of the start of treatment

Exclusion Criteria:

1. Has any one of the following sarcoma sub types: alveolar soft-part sarcoma, chondrosarcoma, dermatofibrosarcoma, Ewing sarcoma, GIST, Kaposi sarcoma, mixed mesodermal tumor, osteosarcoma, radiation induced sarcomas, and unresectable low grade liposarcoma.
2. Clinically evident congestive heart failure >Class II of the New York Heart Association (NYHA) guidelines (Appendix 4)
3. Serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia, or ventricular arrhythmias classified as Lown III, IV, or V (Appendix 4)
4. History and/or signs of active coronary artery disease/ischemia with or without angina pectoris
5. Serious myocardial dysfunction defined as scintigraphically (MUGA [multiple gated acquisition scan], myocardial scintigram) or ultrasound-determined absolute left ventricular ejection fraction (LVEF) <45%
6. History of HIV infection
7. Prior nephrectomy or history of urinary tract obstruction
8. Active, clinically serious infection requiring systemic antibacterial, antifungal, or antiviral therapy
9. Any major surgery within 3 weeks prior to start of treatment
10. Metastatic brain or meningeal tumors, unless the subject is >6 months from definitive therapy and has a negative imaging study within 4 weeks of study entry. In addition, the subject must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable, provided the dose is stable for 1 month prior to study start, and following screening radiographic studies).
11. Previous malignancy (except cervical carcinoma in situ, adequately treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis, & T1] or other malignancies curatively treated >5 years prior to entry)
12. Pregnancy or lactation
13. Substance abuse or medical, psychological, or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
14. Any condition that is unstable or could jeopardize the safety of a subject and his/her compliance with the protocol requirements

    In addition, use of the following therapies and medications-prior or concomitant-would exclude a subject from this study:
15. Anticancer chemotherapy, immunotherapy, or any investigational drug therapy during the study or within 4 weeks of study entry (6 weeks for Mitomycin C)
16. Prior treatment with doxorubicin
17. Radiotherapy within 4 weeks of study entry (palliative radiation to bone lesions is permitted if started or planned prior to Cycle 1, Day 1)
18. Bone marrow transplant or stem cell rescue within 4 months of study entry
19. Growth factors such as G-CSF (granulocyte colony-stimulating factor/filgrastim), or biological response modifiers within 3 weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-08; Primary Completion 2012-04 (Actual); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy analysis will be conducted on the intent-to-treat (ITT) population. All attempts will be made to conduct assessment of disease status every 6 weeks until progression of disease or initiating off protocol anti cancer therapies. | Every 6 weeks until progression

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J Lewis, MD, PhD, Study Director — ZIOPHARM Oncology, Inc
Locations (23):
- United States (18):
  - Santa Monica, California
  - Washington D.C., District of Columbia
  - Tampa, Florida
  - Coeur d'Alene, Idaho
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Iowa City, Iowa
  - Lenaxa, Kansas
  - Albuquerque, New Mexico
  - New York, New York
  - Durham, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- Italy (3):
  - Milan
  - Padua
  - Torino
- Romania (2):
  - Cluj-Napoca
  - Lasi